CLINICAL TRIAL: NCT00992433
Title: A Phase II Study in HIV-seropositive Adults to Assess the Safety and Immunogenicity of an Unadjuvanted Novartis H1N1 Influenza Vaccine Administered at Two Dose Levels
Brief Title: H1N1 Vaccine at Two Dose Levels in HIV Positive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-0073; N01AI80002C
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2011-02

CONDITIONS: Influenza
Keywords: influenza, H1N1, vaccine, human immunodeficiency virus
MeSH Terms: conditions — Influenza, Human; Acquired Immunodeficiency Syndrome

ARMS (2):
- Group 2, 30 mcg (Experimental): CD4<200, n=60; CD4 greater than or equal to 200, n=60. 30 mcg H1N1 vaccine on Day 0 and Day 21.
  Interventions: Biological: Inactivated Influenza H1N1 vaccine
- Group 1, 15 mcg (Experimental): CD4<200, n=60; CD4 greater than or equal to 200, n=60. 15 micrograms (mcg) H1N1 vaccine on Day 0 and Day 21.
  Interventions: Biological: Inactivated Influenza H1N1 vaccine

INTERVENTIONS:
Biological: Inactivated Influenza H1N1 vaccine — Two doses inactivated, licensed, Influenza A (H1N1) 2009 monovalent vaccine; 15 or 30 micrograms (mcg) per dose; slightly opalescent suspension in phosphate buffered saline. 15 mcg dose administered as a single 0.5 mL intramuscular (IM) injection. 30 mcg dose administered as two 0.5 mL IM injections.

SUMMARY:
The purpose of this study is to see how the body reacts to different strengths of the H1N1 flu shot in persons infected with human immunodeficiency virus (HIV). This study will also compare how the CD4 count (cells that help fight disease) affects the body's response to the H1N1 flu shot. In this study, 2 strengths of the H1N1 flu shot will be given twice, about 3 weeks apart. The results of this study will help researchers find out if the different strengths of the H1N1 flu shot make the body produce H1N1 antibodies that are better at fighting H1N1 flu. About 240 HIV positive subjects, ages 18-64 years, will be asked to take part in this study. Study procedures include: blood sampling, physical exams, and use of memory aids to record temperature, medications and symptoms. The length of patient participation is about 7 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization (WHO) to declare a pandemic on June 11, 2009. The immunosuppression associated with human immunodeficiency virus (HIV)-infection has been related to diminished immune responses to vaccination against multiple pathogens, including influenza. The widespread use of antiretroviral therapy has resulted in a significant decrease in the mortality from HIV/acquired immune deficiency syndrome (AIDS) and, as a result, HIV-infected subjects constitute a demographically growing subpopulation in the United States. Currently, novel H1N1 vaccines are being evaluated in the general population. Researchers propose to evaluate the safety and immunogenicity of the novel H1N1 vaccines in HIV-infected subjects, because the data from clinical trials enrolling healthy subjects may not apply to immunosuppressed individuals; and an evaluation of the immune responses to vaccination against new, pandemic influenza viruses has never been performed in HIV-infected subjects. This is a randomized, open label, Phase II study in HIV seropositive males and non-pregnant females, aged 18-64 years. This study is designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine at 2 dose levels. Subjects will be randomized into 2 dose groups, stratified by cluster of differentiation (CD4) cell count at enrollment (120 subjects per dose group with 60 subjects per CD4 cell count stratum, <200/mL or greater than or equal to 200/mL) to receive intramuscular (IM) inactivated influenza H1N1 vaccine at 15 mcg (Group 1) or 30 mcg (Group 2). The H1N1 vaccine will be administered at Day 0 and Day 21. Following immunization, safety will be measured by assessment of adverse events through 21 days following the last vaccination (Day 42 for those receiving both doses and Day 21 for those who do not receive the second dose), serious adverse events and new-onset chronic medical conditions through 7 months post first vaccination (Day 201), and reactogenicity to the vaccine for 8 days following each vaccination (Day 0-7). A CD4/CD8 panel and viral load will be measured prior to first vaccination on Day 0 and at Day 10 post the second vaccination. Immunogenicity testing will include hemagglutination inhibition assay (HAI) and neutralizing antibody testing on serum obtained on the day of each vaccination (prior to vaccination), on Day 10 after each vaccination, 21 days following the second vaccination (Day 42) and 6 months after the second vaccination (Day 201). The primary objectives of this study are: (safety), to assess the safety of the unadjuvanted, inactivated H1N1 vaccine in HIV-1 seropositive adults when administered at the 15 mcg or 30 mcg dose and (immunogenicity) to assess the antibody response following 1 and 2 doses of inactivated H1N1 vaccine administered intramuscularly at the 15 mcg or 30 mcg dose levels in HIV-1 seropositive adults stratified by CD4 count at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus (HIV) infection defined as documented by an enzyme-linked immunosorbent assay (ELISA) and confirmed with a Western blot at any time prior to study entry. Serum HIV-1 antigen, plasma HIV-1 ribonucleic acid (RNA), or any Food and Drug Administration (FDA) approved antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* Males or non-pregnant females age 18-64, inclusive.
* Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, Depo-Provera injections or Implanon implants for at least 30 days following the last vaccination.
* Are medically stable, as determined by the Investigator (based on review of health status, vital signs, medical history, and targeted physical examination. Vital signs must be within normal ranges prior to the first vaccination (heart rate 55-100, blood pressure systolic <160, blood pressure diastolic <90).
* Receipt of the 2009-2010 seasonal influenza vaccine at least two weeks prior to enrollment in this study.
* Intend to be available for follow-up visits and phone call access through 7 months following receipt of H1N1 vaccine.
* Are able to understand and comply with planned study procedures.
* Subject receiving regular medical follow-up care for HIV.
* Has a documented platelet count of >50,000mm^3 and an absolute neutrophil count (ANC) of >500mm^3 within the 3 months prior to study entry.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Treatment for an opportunistic infection (OI) initiated within 2 weeks prior to enrollment, or have symptoms that have not stabilized.
* Have a known allergy to eggs or other components of the vaccine (including polymyxin, neomycin, and chicken protein).
* Women who are pregnant or breastfeeding.
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination.
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have a neoplastic disease that will be treated with chemotherapy or radiation, or a history of any hematologic malignancy.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids. For oral or parenteral: prednisone or equivalent (greater than or equal to 2.0 mg/kg per day or greater than or equal to 20 mg total dose) for more than 2 consecutive weeks (or 2 weeks total) in the past 3 months. For inhaled steroids: >800 mcg/day of beclomethasone dipropionate or equivalent within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have an uncontrolled major psychiatric diagnosis.
* Have a history of receiving immunoglobulin or other blood products within the 3 months prior to vaccination in this study.
* Received an experimental agent (vaccine, drug, biologic, device, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 201 follow-up call).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have a history of severe reactions following previous immunization with influenza virus vaccines.
* Have a moderate-severe acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 72 hours prior to vaccination. (This may result in a temporary delay of vaccination).
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Participated in a novel influenza 2009 H1N1 influenza vaccine study or have history of novel 2009 H1N1 influenza infection prior to enrollment.
* Have a history of alcohol or drug abuse in the last 3 months.
* Plan to travel outside of North America at any time between the first vaccination and 42 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Baltimore - Institute of Human Virology, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] El Sahly HM, Davis C, Kotloff K, Meier J, Winokur PL, Wald A, Johnston C, George SL, Brady RC, Lehmann C, Stokes-Riner A, Keitel WA. Higher antigen content improves the immune response to 2009 H1N1 influenza vaccine in HIV-infected adults: a randomized clinical trial. J Infect Dis. 2012 Mar 1;205(5):703-12. doi: 10.1093/infdis/jir837. Epub 2012 Jan 24. PMID 22275399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were HIV-positive adult males and females recruited from existing patient populations and from the communities at large around the clinical sites. Participants were enrolled between 19Nov2009 and 23Apr2010.
Groups:
- 15 Mcg H1N1 Vaccine: 15 mcg inactivated influenza H1N1 vaccine administered intramuscularly on Day 0 and Day 21.
- 30 Mcg H1N1 Vaccine: 30 mcg inactivated influenza H1N1 vaccine administered intramuscularly on Day 0 and Day 21.
Period: Overall Study
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Started | 95 | 97
Completed | 91 | 90
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine | Total
Number analyzed (Participants) | 95 | 97 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 97 | 192
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (9.9) | 45.3 (9.3) | 45.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 76 | 75 | 151
Region of Enrollment [Number; unit: participants]
  United States | 95 | 97 | 192

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 10 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 10 post first H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 10 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 10 days after the first vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint are included. One participant was excluded due to not meeting eligibility criteria at the time of enrollment. Analyses are as treated. This outcome restricts to CD4 stratum.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 34
Participants | 14 | 23

2. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post first H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 21 days after the first vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 32
Participants | 14 | 21

3. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 10 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 10 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 10 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 10 days after the second vaccination
Population: Participants who received both H1N1 vaccinations in window and from whom blood was collected at the timepoint are included. One participant was excluded due to not meeting eligibility criteria at the time of enrollment. Analyses are as treated. This outcome restricts to CD4 stratum.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 33
Participants | 15 | 23

4. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 21 days after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 32
Participants | 18 | 19

5. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 180 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 180 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 180 days after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 33 | 32
Participants | 9 | 13

6. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 10 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 1
Time Frame: Day 0 prior to vaccination and 10 days after the first vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint are included. Analyses are as treated. This outcome restricts to CD4 stratum.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 58
Participants | 32 | 42

7. Primary Outcome: Number of Participants in the CD4 CD4 200/mL or Greater Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 2
Time Frame: Day 0 prior to vaccination and 21 days after the first vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 58 | 60
Participants | 30 | 42

8. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 10 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 3
Time Frame: Day 0 prior to vaccination and 10 days after the second vaccination
Population: Participants who received both H1N1 vaccinations in window and from whom blood was collected at the timepoint are included. Analyses are as treated. This outcome restricts to CD4 stratum.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 55 | 57
Participants | 32 | 41

9. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 4
Time Frame: Day 0 prior to vaccination and 21 days after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 55 | 57
Participants | 30 | 40

10. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With 4-Fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 5
Time Frame: Day 0 prior to vaccination and 180 days after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 54 | 55
Participants | 16 | 27

11. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus at Baseline and 10 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants at Day 0 prior to vaccination and 10 days after the first vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 0 prior to vaccination and 10 days after the first vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 34
Participants
  Day 0 | 7 | 8
  Day 10 | 16 | 24

12. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after the first vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the first vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 32
Participants | 16 | 22

13. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 10 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 10 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 10 after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 33
Participants | 17 | 24

14. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 34 | 32
Participants | 20 | 22

15. Primary Outcome: Number of Participants in the CD4 Less Than 200/mL Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 180 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 180 after the second vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 33 | 32
Participants | 12 | 19

16. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus at Baseline Prior to the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants at Day 0 prior to the first vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 0 prior to the first vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 61
Participants | 11 | 11

17. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 10 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants 10 days after the first vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 10 after the first vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 60 | 58
Participants | 40 | 45

18. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 12
Time Frame: Day 21 after the first vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 58 | 60
Participants | 37 | 45

19. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 10 and 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 10 and 21 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 10 and Day 21 after the second vaccination
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 55 | 57
Participants
  Day 10 Post Second Dose | 38 | 43
  Day 21 Post Second Dose | 36 | 42

20. Primary Outcome: Number of Participants in the CD4 200/mL or Greater Stratum With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 15
Time Frame: Day 180 after the second vaccination
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 54 | 55
Participants | 25 | 32

21. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, and nausea for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days post first vaccination (Day 0-7).
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 97
Participants
  Feverishness | 11 | 6
  Malaise | 22 | 20
  Myalgia | 14 | 20
  Headache | 24 | 26
  Nausea | 12 | 9

22. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 21
Time Frame: Within 8 days post second vaccination (Day 0-7).
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 89 | 94
Participants
  Feverishness | 8 | 10
  Malaise | 14 | 14
  Myalgia | 14 | 14
  Headache | 11 | 20
  Nausea | 7 | 9

23. Primary Outcome: Number of Participants Reporting Fever After the First Vaccination
Description: Participants were provided a thermometer and a memory aid to record daily oral temperatures for 8 days (Day 0-7) after vaccination. Participants are counted as experiencing fever if they reported oral temperatures of 38 degrees Celsius or higher on any of the 8 days.
Time Frame: Within 8 days post first vaccination (Day 0-7).
Population: Participants who received the first vaccination are included. One participant did not record temperatures. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 96
Participants | 0 | 1

24. Primary Outcome: Number of Participants Reporting Fever After the Second Vaccination
Description: as for outcome 23
Time Frame: Within 8 days post second vaccination (Day 0-7).
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 89 | 94
Participants | 1 | 2

25. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days post first vaccination (Day 0-7).
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 97
Participants
  Pain | 14 | 22
  Tenderness | 19 | 31
  Swelling | 9 | 7

26. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the Second Vaccination
Description: as for outcome 25
Time Frame: Within 8 days post second vaccination (Day 0-7).
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 89 | 94
Participants
  Pain | 8 | 16
  Tenderness | 11 | 25
  Swelling | 8 | 6

27. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Within 8 days post first vaccination (Day 0-7).
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 97
Participants
  Redness | 12 | 13
  Swelling | 9 | 7

28. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the Second Vaccination
Description: as for outcome 27
Time Frame: Within 8 days post second vaccination (Day 0-7).
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 89 | 94
Participants
  Redness | 12 | 8
  Swelling | 9 | 6

29. Primary Outcome: Number of Participants Reporting Vaccine-Associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; may have jeopardized the participant or required intervention to prevent one of these outcomes; or was described as Guillain-Barré Syndrome. Association to vaccination was determined by a study clinician licensed to make medical diagnosis.
Time Frame: Day 0 through Day 180 after the last vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 97
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | 15 Mcg H1N1 Vaccine | 30 Mcg H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 8/95 | 5/97
Other Adverse Events (participants affected / at risk) | 61/95 | 73/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 Mcg H1N1 Vaccine (N=95) | 30 Mcg H1N1 Vaccine (N=97)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 Mcg H1N1 Vaccine (N=95) | 30 Mcg H1N1 Vaccine (N=97)
Blood pressure increased (Investigations) | 8 (8) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 8 (10)
Feeling hot (General disorders) | 14 (19) | 14 (16)
Malaise (General disorders) | 25 (36) | 28 (34)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (28) | 24 (34)
Headache (Nervous system disorders) | 29 (35) | 33 (46)
Nausea (Gastrointestinal disorders) | 17 (19) | 13 (18)
Injection site pain (General disorders) | 18 (22) | 30 (38)
Tenderness (General disorders) | 25 (30) | 41 (56) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 16 (24) | 17 (21)
Injection site swelling (functional grading) (General disorders) | 13 (17) | 10 (13) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 14 (18) | 10 (13) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less